CLINICAL TRIAL: NCT01258309
Title: Safety and Efficacy of Olopatadine Hydrochloride/Ketorolac Tromethamine Ophthalmic Solution Compared With Olopatadine Hydrochloride Ophthalmic Solution in Patients With Seasonal Allergic Conjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Olo-keto/2009
Record Dates: First submitted 2010-12-09; First posted 2010-12-10 (Estimated); Last update posted 2012-01-25 (Estimated); Status verified 2012-01

CONDITIONS: Rhinitis, Allergic, Seasonal; Conjunctivitis, Allergic
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Conjunctivitis, Allergic | interventions — Olopatadine Hydrochloride; Ketorolac Tromethamine; Ophthalmic Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): olopatadine hydrochloride/ketorolac tromethamine fixed dose combination ophthalmic solution
  Interventions: Drug: olopatadine hydrochloride /ketorolac tromethamine fixed dose combination ophthalmic solution
- 2 (Active Comparator): olopatadine hydrochloride/ketorolac tromethamine fixed dose combination ophthalmic solution
  Interventions: Drug: olopatadine hydrochloride 0.1% ophthalmic solution

INTERVENTIONS:
Drug: olopatadine hydrochloride /ketorolac tromethamine fixed dose combination ophthalmic solution — One drop of olopatadine hydrochloride/ketorolac tromethamine fixed dose combination ophthalmic solution administered to each eye, twice daily for 21 days.
  Arms: 1
Drug: olopatadine hydrochloride 0.1% ophthalmic solution — One drop of olopatadine hydrochloride 0.1% ophthalmic solution administered to each eye, twice daily for 21 days.
  Other Names: Patanol®
  Arms: 2

SUMMARY:
This study will investigate the safety and efficacy of olopatadine hydrochloride / ketorolac tromethamine fixed dose combination ophthalmic solution compared with olopatadine hydrochloride ophthalmic solution in patients with seasonal allergic conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of seasonal allergic conjunctivitis

Exclusion Criteria:

* Ocular infection or history of ocular herpes infection
* History of retinal detachment or diabetic retinopathy
* Prior or current use of systemic or topical steroids, NSAIDs, anticholinergics, immunosuppressants, or antihistamines
* Ocular surgery within 8 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2010-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Ocular Itching | Day 21

SECONDARY OUTCOMES:
Hyperemia | Day 21
Chemosis | Day 21
Ocular mucous discharge | Day 21

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Bangalore, Karnataka, India